CLINICAL TRIAL: NCT01241799
Title: A Prospective, Single Blinded, Randomized, Controlled Study to Compare the Yield of Endoscopic Ultrasound Guided Fine Needle Aspiration (EUS-FNA) With and Without the Use of a Stylet in the Biopsy Needle
Brief Title: Yield of Endoscopic Ultrasound Guided Fine Needle Aspiration (EUS-FNA) With and Without the Use of a Stylet in the Biopsy Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Eric Lam, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: H08-01481
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Pancreatic Mass on Imaging
Keywords: endoscopic ultrasound guided fine needle aspiration (EUS-FNA); pancreatic biopsy; randomized; single blind; fine needle aspiration (FNA) adequacy; fine needle aspiration (FNA) accuracy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Pancreatic biopsy with stylet in then stylet out
  Interventions: Procedure: Endoscopic ultrasound guided fine needle aspiration biopsy
- 2 (Experimental): Pancreatic biopsy with stylet out then stylet in
  Interventions: Procedure: Stylet out FNA first, Stylet in FNA second

INTERVENTIONS:
Procedure: Endoscopic ultrasound guided fine needle aspiration biopsy — 22 gauge fine needle aspiration biopsy of the pancreatic mass with the stylet in. Vacuum suction applied. 12 intra mass needle passes done. A new 22 gauge FNA biopsy needle with the style out is then used to biopsy the pancreatic mass. Vacuum suction applied. 12 intra mass needle masses done.
  Arms: 1
Procedure: Stylet out FNA first, Stylet in FNA second — 22 gauge FNA biopsy of pancreatic mass with the stylet out. Vacuum suction applied. 12 intra mass needle passes done. A new 22 gauge FNA biopsy needle with the stylet in is used to biopsy the pancreatic mass. Vacuum suction applied. 12 intra mass needle passes done.
  Arms: 2

SUMMARY:
Purpose:

To compare the diagnostic yield of endoscopic ultrasound guided fine needle aspiration biopsy (EUS-FNA) in patient with pancreatic masses with and without the use of a stylet in place within the biopsy needle.

Hypothesis:

In patients undergoing an EUS FNA for pancreatic indications, patients having a fine needle aspiration biopsy (FNA) without the internal stylet will have a greater diagnostic yield compared to those with the internal stylet.

Justification:

EUS-FNA is an increasingly important means of obtaining tissue samples from lesions within the thorax and abdomen. In experienced hands EUS-FNA is a safe alternative to more invasive procedures such as mediastinoscopy or laparoscopy. EUS-FNA can be used for sampling suspected cholangiocarcinoma, pancreatic masses or cysts, submucosal gastric lesions, peripancreatic, perigastric or mediastinal lymph nodes and in some cases adrenal or liver masses. Therefore, it is a powerful tool for both diagnosis and tumour staging. For example, for the diagnosis of pancreatic adenocarcinoma, which is a common indication for EUS-FNA, the sensitivity varies from 75 to >90%, with a specificity of 82-100% and a mean accuracy of 85%. Improving the diagnostic yield may lead to an earlier diagnosis with a reduced number of investigations and earlier institution of treatment for the patient.

The FNA needle system consists of a 22 or 19 gauge needle which is manipulated by a handle piston that attaches to the biopsy channel of the endoscopic ultrasound (EUS) linear scope. The tip of the needle has grooves to disperse ultrasound waves making the tip of the needle easily seen. The sample is taken by inserting a specially designed needle into the area of interest under EUS guidance. Inside the needle is a removable stylet with a rounded or bevelled tip to facilitate the passage of the needle into the tissue. The usual practice is for the stylet to be extracted after the needle has been passed into its optimum position within the tissue and for it to be re-inserted before each pass. However, a recent prospective trial with 111 patients, published in abstract form, found this approach was associated with a significant reduction in the proportion of adequate samples compared to when the stylet was removed before passing the needle. Although there was no significant difference in the diagnostic yield between the two groups this study raises the issue that the stylet left in place is to the detriment of the tissue sample and, ultimately, may reduce the diagnostic yield or increase the number of passes needed to obtain a satisfactory sample.

One limitation to this study includes the heterogenous patient population. Yields of EUS-FNA vary considerably depending on the type of tissue being biopsied. The second limitation is that consecutive patients were randomized to having the stylet removed versus having the stylet not removed at the time of FNA. There is no control group from which to compare the two groups. An improvement in the study design would be to have each patient to be their own control group. Successive passes of the FNA needle can increase the bloodiness of the sample, so randomization of the order in which each group is done will help eliminate potential bias.

It is clear from the current published literature that removing the stylet increases the cellularity of the sample. However, this increased cellularity may be the result of more contamination from the GI tract through which the FNA needle needs to pass in order to get an extra-luminal sample. Blood or a traumatic FNA can also lead to increased cellularity that can compromise diagnostic accuracy.

Diagnostic yield depends on both adequacy of the sample and enough cells from the lesion to interpret. A preliminary result based on an air dried slide often can lead to fewer FNA passes if a diagnosis can be made. If this is not possible, a cell block preparation is made from all the washings from the EUS-FNA needle. No study has examined the diagnostic accuracy of these two types of samples using an EUS-FNA needle with and without the stylet within the same patient.

Objectives:

To determine if the diagnostic yield of EUS-FNA is increased if the stylet is removed from the FNA needle compared with leaving it in place.

DETAILED DESCRIPTION:
Research Method:

All patients referred for EUS who are also likely to require FNA will be screened for study eligibility by way of the inclusion and exclusion criteria. After informed consent has been obtained patients will be randomized to 2 different groups by random number generation

1. Stylet in FNA first, Stylet out FNA second
2. Stylet out FNA first, Stylet in FNA second As each method of tissue sampling will be used for all patients they will effectively act as their own controls.

In patients randomized to the first group the stylet in is left in place within the needle for the first three passes of the needle into the area to be sampled. A new 22 gauge EUS FNA is then used to obtain the FNA with the stylet out.

In patients randomized to the second group a 22 gauge EUS FNA needle with the stylet out is used for the first three passes. A new needle with the stylet in is subsequently used for further sampling. Three passes will be done for each FNA biopsy.

For each patient the sample adequacy, the number of bloody passes and the number of passes required to obtain an adequate sample will be recorded by the cytopathology technician. Each tissue sample will be prepared and analysed by experienced on-site cytopathology staff, who will be blinded to the group allocation of the respective patients. A positive or negative diagnosis will be recorded when the final cytology result is available. At the end of the study period a comparison between the two groups will be made in relation to the parameters outlined above.

Statistical Analysis:

Endpoints:

The primary endpoint of our study will be the number of samples with a positive diagnosis in each group. Secondary end-points will be the number of bloody passes, the sample adequacy and the number of passes needed to obtain an adequate sample.

Sample size calculation:

The outcome will be represented as a proportion of FNA samples that have a positive diagnosis. The effect size between the stylet in FNA and stylet out FNA is expected to be 30%. This is at a significance level of p= 0.05 and 80% power. The number of patients in each arm is therefore 36.

Description of methodology All patients who are referred for a pancreatic EUS and are likely to require an FNA will be identified and screened for eligibility for entry into the study according to the inclusion and exclusion criteria. Those patients who are seen in the office prior to an EUS appointment will be invited to enter the study by a research nurse or research assistant not involved with the procedure. They will be provided with written and verbal information on the study prior to making their decision. For patients who are referred directly for an EUS-FNA from another physician and who are not seen in the office beforehand a written invitation to enter the study will be sent in advance. This will provide detailed information on the research proposal as well as a helpline number which patients can use to contact one of the study co-ordinators for further advice. A follow up phone call to patients will be made by a study co-ordinator before they attend for the EUS; the initial contact letter will outline when this call will be made, and by whom.

If patients elect to enter into the study informed consent will be obtained prior to randomization.

Summary of procedures In patients randomized to the first group, under intravenous sedation, a linear endoscopic ultrasound examination is performed. The pancreatic mass is identified by endoscopic ultrasound and using a 22 gauge EUS FNA needle with the stylet in is used for the first pass. The stylet is then withdrawn and 10cc of suction is applied to the FNA needle. A sample is obtained by moving the needle in and out of the lesion for a minimum of 15 times. The sample is then collected for cytopathology. The stylet is replaced in the needle and another pass is performed by the same technique. Three passes will be done for each FNA biopsy. A new 22 gauge EUS FNA is then used to obtain the FNA with the stylet out by the same technique as outlined above.

In patients randomized to the second group, under intravenous sedation a linear endoscopic ultrasound examination is performed. The pancreatic mass is identified by endoscopic ultrasound and using a 22 gauge EUS FNA needle with the stylet out is used for the first pass. The stylet is then withdrawn and 10cc of suction is applied to the FNA needle. A sample is obtained by moving the needle in and out of the lesion for a minimum of 15 times. The sample is then collected for cytopathology. The stylet is replaced in the needle and once loaded into position, the stylet is removed prior to starting another pass performed by the same technique. Three passes will be done for each FNA biopsy.

Adverse events that can potentially occur include oversedation (1:500), pancreatitis (1:1000), perforation (1:5000), and bleeding (extremely rare with only one reported case in press) For each patient the sample adequacy, the number of bloody passes and the number of passes required to obtain an adequate sample will be recorded by the cytopathology technician. Each tissue sample will be prepared and analysed by experienced on-site cytopathology staff, who will be blinded to the group allocation of the respective patients. A positive or negative diagnosis will be recorded when the final cytology result is available. At the end of the study period a comparison between the two groups will be made in relation to the parameters outlined above.

Follow-up:

Within one day, all patients will be contacted to determine if any adverse events have occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 19 years of age and older
2. Patients undergoing EUS FNA for solid lesions in the pancreas

Exclusion Criteria:

1. Pancreatic cystic lesions without significant mass effect
2. Pancreatic masses that cannot be accessed by transduodenal FNA in surgically resectable cases
3. Known chronic pancreatitis with pancreaticolithiasis
4. History of acute pancreatitis in the preceding 4 weeks
5. History of gastric surgery or symptoms of gastric outlet obstruction
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of our study will be the number of samples with a positive diagnosis in each group | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lam, Dr., Principal Investigator — University of British Columbia; Jennifer Telford, Dr., Study Director — University of British Columbia; Mark McLoughlin, Dr., Study Director — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada